CLINICAL TRIAL: NCT05453565
Title: Fluid Restricted Resuscitation in Sepsis With Hypotension Meta-Analysis (FRESHLY): Individual Patient Data Met-analysis of the ARISE FLUIDS, CLASSIC, CLOVERS and EVIS Trials
Brief Title: Restricted or Liberal Fluid for Haemodynamic Resuscitation in Sepsis
Acronym: FRESHLY
Status: Not yet recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: FRESHLY V1
Record Dates: First submitted 2022-06-03; First posted 2022-07-12 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Septic Shock; Fluid Resuscitation
MeSH Terms: conditions — Shock, Septic | interventions — Vasoconstrictor Agents; Fluid Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vasopressors: A haemodynamic resuscitation strategy based upon the restriction of IV fluids (by either volume or rate of infusion) with initiation or change of rate of vasopressors if required to meet perfusion targets
  Interventions: Other: Vasopressors
- Fluids: A strategy of resuscitation with intravenous fluids as the primary intervention to achieve perfusion targets with subsequent initiation or change of rate of vasopressors if required.
  Interventions: Other: Fluids

INTERVENTIONS:
Other: Vasopressors — A haemodynamic resuscitation strategy based upon the restriction of IV fluids (by either volume or rate of infusion) with initiation or change of rate of vasopressors if required to meet perfusion targets
  Groups: Vasopressors
Other: Fluids — A strategy of resuscitation with intravenous fluids as the primary intervention to achieve perfusion targets with subsequent initiation or change of rate of vasopressors if required.
  Groups: Fluids

SUMMARY:
A prospective, individual patient data meta-analysis (IPDMA) of four multicentre, open-label, randomised clinical trials of initial haemodynamic resuscitation in patients with septic shock.

DETAILED DESCRIPTION:
This study is a prospective, individual patient data meta-analysis (IPDMA) of four multicentre, open-label, randomised clinical trials of initial haemodynamic resuscitation in patients with septic shock.

The investigators will include four multicentre, open-label, randomised, clinical trials:

* Australasian Resuscitation in Sepsis Evaluation Fluids of Vasopressors in Emergency Department Sepsis (ARISE FLUIDS) trial conducted in Australia and New Zealand. ClinicalTrials.gov identifier NCT04569942
* Conservative versus Liberal Approach to fluid therapy of Septic Shock in intensive Care (CLASSIC) trial conducted in seven European countries. ClinicalTrials.gov identifier NCT03668236
* Crystalloid Liberal or Vasopressors Early (CLOVERS) trial conducted in the United States. ClinicalTrials.gov identifier NCT03434028
* Early Vasopressors in Sepsis (EVIS) trial conducted in the United Kingdom. ClinicalTrials.gov identifier NCT05179499

All four trials have all received relevant approval from a research ethics committee with a locally appropriate method of obtaining consent. These trials are prospectively chosen prior to the results of any individual trial being known because they are investigating the same broad question in patients with acute septic shock across several countries. The investigators of these trials collaborated to harmonise data and outcomes as far as possible across all trials to facilitate an IPDMA.

The aims to provide high level evidence to address the question of whether a fluid sparing/early vasopressor approach or a liberal fluid/later vasopressor approach to initial haemodynamic resuscitation in septic shock results in improved outcomes, including mortality.

ELIGIBILITY:
Inclusion Criteria:

Participants of the ARISE FLUIDS, CLASSIC, CLOVERS & EVIS trials who had:

* Suspected or proven infection
* Systolic blood pressure (SBP) <100 mm Hg OR mean arterial pressure (MAP) <65 mm Hg
* Lactate ≥ 2.0 mmol/L
* Requirement for vasopressors to meet perfusion targets

Exclusion criteria:

Participants not in the ARISE FLUIDS, CLASSIC, CLOVERS & EVIS trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trials include adult patients requiring resuscitation for hypotension or hypoperfusion due to suspected sepsis as defined in the original studies. Participants may be enrolled in the emergency department, acute care ward or intensive care unit.
Sampling Method: Probability Sample
Enrollment: 7838 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 days post randomisation | 90 days
  Death from any cause at 90 days after randomisation

SECONDARY OUTCOMES:
Time from randomisation to death | Up to day 90
  Time from randomisation to death
Incidence of mechanical ventilation | from randomisation until day 90 post-randomisation
  Commencement of mechanical ventilation from randomisation until day 90 post-randomisation
Incidence of acute renal replacement therapy | from randomisation until day 90 post-randomisation
  Commencement of renal replacement therapy from randomisation until day 90 post-randomisation
Days alive free of organ support at 28 days post randomisation | from randomisation until day 28 post-randomisation
  days the patient is alive and receiving nil organ support from from randomisation until day 28 post-randomisation
Duration of hospital stay | From randomisation until day 90 post-randomisation
  Length of time in hospital from randomisation until death or hospital discharge or day 90 post-randomisation
Incidence of serious adverse events | from randomisation until day 90 post-randomisation
  Number of adverse events from randomisation until day 90 post-randomisation
Duration of intensive care unit (ICU) stay | From randomisation until day 90 post-randomisation
  Length of time in ICU from randomisation until death or hospital discharge or day 90 post-randomisation